CLINICAL TRIAL: NCT04057599
Title: Investigation of Postoperative Ileus After Lumbar Spine Surgery: a Prospective Observational Study
Brief Title: Ileus After Lumbar Spine Surgery
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907033RINB
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2019-08

CONDITIONS: Lumbar Spine Surgery Postoperative Ileus
Keywords: post-operative ileus,lumbar spine surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative ileus (POI) after lumbar spine surgery is not uncommon. However, the incidence, severity and risk factors of ileus after spine surgery remain uncertain because there is not yet a prospective investigation using a subjective grading evaluation tool.

DETAILED DESCRIPTION:
This study aims to prospectively investigate the incidence of POI after spine surgery by using the I-FEED scoring system. The severity of POI after spine surgery thus could be stratified and then an investigation of possible risk factors could be identified.

ELIGIBILITY:
Adult patients who undergoing elective lumbar spine surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergoing elective lumbar spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2019-08-17 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Validation of the I-FEED scoring system | 3 days
  Construct validation of the I-FEED scoring system to ileus-related outcome including the need of gastrointestinal medication, the length of hospital stay and in-hospital cost

CONTACTS AND LOCATIONS:
Overall Officials: Fon-Yih Tsuang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan